CLINICAL TRIAL: NCT06795750
Title: The Effect of Neural Therapy on Heart Rate Recovery, Cardiac Parameters and Pain in Fibromyalgia: a Randomized Controlled Trial
Brief Title: The Effect of Neural Therapy on Heart Rate Recovery, Cardiac Parameters and Pain in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Sebahat Tekeli Sengul, assistant professor, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sengul-UsakU
Record Dates: First submitted 2025-01-03; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia Syndrome
Keywords: neural therapy; fibromyalgia; autonomic dysfunction
MeSH Terms: conditions — Fibromyalgia; Primary Dysautonomias | interventions — Anesthesia, Local; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- neural therapy and exercise (Experimental): The neural therapy group received local injections of 1% lidocaine into the C5-L2 segmental and painful points once a week for 5 weeks.
  Interventions: Procedure: neural therapy
- exercise (Experimental): The second group received a home exercise programe consisting of stretching, strengthening, and aerobic exercises for 30 minutes, three times per week, for a duration of five weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Procedure: neural therapy — Neural therapy (NT) is a therapeutic intervention that uses local anesthetics to alleviate persistent musculoskeletal pain. NT targets the underlying autonomic dysfunction by modulating the autonomic nervous system. The enhancement of autonomic dysfunction leads to controlled microcirculation, the elimination of pain mediators, and the attainment of an anti-inflammatory effect. NT focuses on painful regions, specific segments of these areas, and trigger points, encompassing both local and segmental treatment
  Arms: neural therapy and exercise
Other: Exercise — The second group received a home exercise program consisting of stretching, strengthening, and aerobic exercises for 30 minutes, three times per week, for a duration of five weeks.
  Arms: exercise

SUMMARY:
Background: Autonomic dysfunction has been observed in patients with fibromyalgia and is associated with symptoms and arrhythmia development in such patients.The investigators can analyze dysautonomia using heart rate recovery (HRR). Studies have reported that impaired HRR improves after exercise in fibromyalgia patients. Although previous theories have suggested that neural therapy benefits fibromyalgia patients by regulating autonomic dysfunction, there are no studies in the literature reporting that neural therapy improves autonomic dysfunction.

Aims: The purpose of the present study was to compare whether neural therapy + exercise therapy provided more improvement in impaired HRR, cardiac parameters, and pain levels than exercise alone therapy in fibromyalgia patients with autonomic dysfunction.

Methods: The study included sixty female patients diagnosed with fibromyalgia and impaired HRR, all over the age of 18. The investigators divided the patients into two groups: the exercise-alone group and the neural therapy + exercise group.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic condition characterized by musculoskeletal pain, exhaustion, sleep disturbances, and tenderness at specific trigger points in the musculoskeletal system. The frequency of fibromyalgia syndrome (FMS) varies between 3% and 6%, with more frequent detection in women. Dysautonomia, a form of autonomic nervous system dysfunction, is present in one-third of patients with fibromyalgia. The heart rate recovery index and/or the head-up tilt table test can diagnose dysautonomia. It may play a central role in the pathogenesis of the disease and explain multiple systemic symptoms.

The investigators calculate heart rate recovery (HRR) by subtracting the heart rate at the 30th second or 1st, 2nd, 3rd, 4th, 5th, and 10th minutes during the post-exercise recovery period from the maximum heart rate during the treadmill exercise test. The investigators see an abnormal HRR index as a sign of autonomic dysfunction, primarily cardiovascular disease, and as a predictor of all-cause mortality, including cardiovascular mortality.

Neural therapy (NT) is a therapeutic intervention that uses local anesthetics to alleviate persistent musculoskeletal pain. NT targets the underlying autonomic dysfunction by changing the autonomic nervous system. This controls microcirculation, gets rid of pain mediators, and reduces inflammation. Numerous European countries, particularly Germany, have used NT, but studies on its effectiveness in fibromyalgia patients are scarce. The present study aims to investigate whether neural therapy improves cardiac parameters and autonomic dysfunction in fibromyalgia patients with dysautonomia and its effect on pain.

The study included sixty female patients diagnosed with fibromyalgia and impaired HRR, all over the age of 18. İnvestigators divided the patients into two groups: the exercise alone group and the neural therapy + exercise group.The study involved patients diagnosed with fibromyalgia who were over 18 years old and consented to participate in neural and exercise therapy. The investigators excluded from the study patients with conditions that could induce secondary fibromyalgia syndrome, rheumatic diseases, infectious diseases, neurological disorders, allergies to lidocaine, infections, open wounds, vascular pathologies, severe systemic illnesses, significant mental disorders, or serious psychiatric conditions. The study also excluded smokers, alcoholics, individuals with known cardiovascular, respiratory, or neurological disorders or musculoskeletal injuries, and those participating in regular competition or individual sports.

The study used a stress ECG test, the Bruce Protocol-based maximum treadmill stress test, to identify patients with significant autonomic dysfunction. The investigators recorded heart rate, systolic blood pressure, and diastolic blood pressure after a 15-minute rest period. The volunteers then exercised on a treadmill at a speed of 5 km/h and 1% incline for the first 5 minutes of warm-up and at the same incline until they reached the maximum heart rate. İnvestigators recorded HR, SBP, and DBP on the 1st, 2nd, 3rd, 4th, 5th, and every 5 minutes until the end of the rest period.

The study divided the group whose HRR decreased by less than 12 beats in the 1st minute and less than 22 beats in the 2nd minute into neural therapy + exercise and exercise alone groups using the closed envelope method. The neural therapy group underwent neural therapy for five weeks at one-week intervals, while the exercise group engaged in a 30-minute home exercise program three times a week for the same duration.

The investigators examined HRR changes, VAS scores, and cardiac parameters in both groups before and after treatment. The investigators investigated whether there was a significant difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

-Clinical diagnosis of Fibromiyalgia Syndrome

Exclusion Criteria:

* Secondary fibromyalgia syndrome (such as systemic lupus erythematosus, scleroderma, and Sjögren syndrome), those suffering from rheumatic diseases like polymyalgia rheumatica
* Infectious diseases
* Neurological disorders including thyroid dysfunction, neuropathies, myopathies, myositis, and multiple sclerosis
* Allergies to lidocaine and its constituents -Infections, open wounds, or vascular pathologies at the site of application -
* Severe systemic illnesses Significant mental disorders, or serious psychiatric conditions
* Malignancies or anticoaglant usage
* Pregnancies and breastfeeding experiences
* Who underwent physical therapy, rehabilitation, or injection therapy within the last six months
* Smokers (as they might affect the heart rate recovery index),
* alcoholics
* who did regular individual sports

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in impaired heart rate recovery | From enrollment to the end of treatment at 5 weeks
  Heart rate recovery (HRR) can be calculated by subtracting the heart rate at the 30th second or 1st, 2nd, 3rd, 4th, 5th, and 10th minutes during the post-exercise recovery period from the maximum heart rate during the treadmill exercise test (the most commonly used is the 1st minute [HRR60 s] and the 2nd minute [HRR120]). An abnormal HRR index was defined as a drop in the heart rate of less than 12 beats in the first minute and 22 beats in the second minute during the resting period (HRR60 s <12) (HRR120 s <22).

SECONDARY OUTCOMES:
Changes in pain levels in fibromiyalgia patients | From enrollment to the end of treatment at 5 weeks
  The pain level was assessed with the Visual Analog Scale (VAS) using a 10-cm ruler. All patients were told that no pain corresponded to 0, the most severe pain to 10, and moderate pain to five points and asked to describe their pain accordingly.
Changes in heart rate | From enrollment to the end of treatment at 5 weeks
  Heart rate number of cardiac cycles in beats per min.
Changes in blood pressure | From enrollment to the end of treatment at 5 weeks
  BP measurement was performed using the Omron HEM 907 oscillometric monitor (Omron Healthcare) with a cuff size appropriate for the arm. The monitor was programmed such that the cuff did not start to inflate until the participant rested quietly for 5 minutes in a seated position with the arm at the level of the heart.

CONTACTS AND LOCATIONS:
Overall Officials: professor, Principal Investigator — Uşak University
Locations (1):
- Faculty of Medicine Department of Cardiology, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No